CLINICAL TRIAL: NCT01473589
Title: Effect of Teriparatide on Femoral Neck Fracture Healing
Brief Title: Effect of Teriparatide on Hip Fracture Healing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13467; B3D-MC-GHDN (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Femur Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Administered once daily by subcutaneous (SC) injection for 6 months
  Interventions: Drug: Placebo; Dietary Supplement: Calcium supplementation; Dietary Supplement: Vitamin D supplementation
- Teriparatide (Experimental): 20 microgram (µg) administered once daily by SC injection for 6 months
  Interventions: Drug: Teriparatide; Dietary Supplement: Calcium supplementation; Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Drug: Teriparatide — Administered by SC injection
  Other Names: Forteo; Forsteo; LY333334
  Arms: Teriparatide
Drug: Placebo — Administered by SC injection
  Arms: Placebo
Dietary Supplement: Calcium supplementation — Administered orally
Dietary Supplement: Vitamin D supplementation — Administered orally

SUMMARY:
The purpose of this study is to see whether teriparatide, given for 6 months versus placebo, will improve the healing of hip (femoral neck) fractures that are repaired during surgery using certain types of orthopedic screws. The study will enroll men and postmenopausal women at least 50 years of age with a recent hip (femoral neck) fracture caused by low-trauma (for example, fall from standing height or less).

DETAILED DESCRIPTION:
This is a 12-month, Phase 3, prospective, randomized, parallel, double-blind, placebo-controlled, multicenter, multinational study to evaluate the effect of 6 months of treatment with teriparatide on fracture healing in participants who have sustained a recent low-trauma, unilateral, femoral neck fracture stabilized by internal fixation. The study has 3 periods:

1. A screening period that must be completed in ≤ 14 days after operative treatment of the femoral neck fracture
2. A 6-month double-blind treatment period [teriparatide 20 µg or placebo given once daily by SC injection]
3. A 6-month observation period.

The primary objective is to assess the effect of 6 months of treatment with teriparatide 20 µg/day versus placebo on the proportion of men and postmenopausal women of at least 50 years of age with no revision surgery 12 months after internal fixation of a low-trauma femoral neck fracture.

All participants will receive supplements of calcium and vitamin D beginning at screening and continuing for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and postmenopausal women who were ambulatory before sustaining a low-trauma, unilateral femoral neck fracture (displaced or nondisplaced)
* Other than femoral neck fracture, be free of incapacitating conditions and have a life expectancy of at least 2 years
* Have received or are eligible for treatment with internal fixation (sliding hip screw or multiple cancellous screws) for the femoral neck fracture (the surgical procedure itself is not performed as part of this study)
* Have given written informed consent (participant or proxy) after being informed of the risks, medications, and study procedures

Exclusion Criteria:

* Increased baseline risk of osteosarcoma
* History of unresolved skeletal diseases affecting bone metabolism other than primary osteoporosis
* Abnormally elevated serum calcium at screening
* Abnormally elevated serum intact parathyroid hormone (PTH) (1-84) at screening
* Severe vitamin D deficiency at screening
* Active liver disease or jaundice
* Significantly impaired renal function
* Abnormal thyroid function not corrected by therapy
* History of malignant neoplasm in the 5 years prior to screening
* History of bone marrow or solid organ transplantation
* History of symptomatic nephrolithiasis or urolithiasis in the 1 year prior to screening
* Previous treatment with the following bone active drugs is allowed but must be discontinued at screening: oral bisphosphonates, selective estrogen receptor modulators (SERMs), calcitonin, estrogen (oral, transdermal, or injectable), progestin, estrogen analog, estrogen agonist, estrogen antagonist or tibolone, and active vitamin D3 analogs. Androgen or other anabolic steroid use must be discontinued, except for use of physiologic replacement testosterone
* Previous treatment with the following bone active drugs is exclusionary, if the stated treatment durations have been met: strontium ranelate for any duration, intravenous bisphosphonates in the 12 months preceding screening, and/or denosumab in the 6 months preceding screening
* Prior treatment with PTH, teriparatide, or other PTH analogs, or prior participation in any other clinical trial studying PTH, teriparatide, or other PTH analogs
* Local or systemic treatment with bone morphogenic proteins or any other growth factor
* Previous fracture(s) or bone surgery in the currently fractured hip
* Soft-tissue infection at the operation site
* Treatment with bone grafting or osteotomies
* Treatment with augmentation using any type of degradable cement, hydroxyapatite-coated implants, or with noninvasive interventions
* Associated major injuries of a lower extremity including fractures of the foot, ankle, tibia, fibula, knee, femur, femoral head or pelvis; dislocations of the ankle, knee or hip

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (91):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laguna Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., York, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Penrith, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Albans, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newmarket, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Catharines, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Jérôme, Quebec
- Denmark (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aarhus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hillerød
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Koege
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tartu, Estonia
- Finland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hong Kong, Hong Kong
- India (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Attavar, Mangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagpur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vadodara
- Israel (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
- Japan (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ohita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shimane
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyko
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamanashi
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga, Latvia
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- New Zealand (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christchurch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takapuna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington South
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tønsberg, Norway
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marbella
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mölndal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Teriparatide 20 micrograms (µg) administered once-daily by subcutaneous (SC) injection for 6 months. Participants received calcium and vitamin D supplements.
- Placebo: Placebo administered once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
Period: Overall Study
Arm/Group | Teriparatide | Placebo
Started | 60 | 62
Received at Least 1 Dose of Study Drug | 60 (Randomized participants who received at least 1 dose of study drug.) | 61 (Randomized participants who received at least 1 dose of study drug.)
Completed 6 Months | 51 | 54
Completed 12 Months | 49 | 48
Completed | 49 | 46
Not Completed | 11 | 16
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 11
Not completed — Physician Decision | 0 | 1
Not completed — Entry criteria not met | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study drug.
Groups:
- Teriparatide: Teriparatide 20 µg administered once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.49 (11.321) | 70.96 (12.023) | 69.73 (11.698)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 34 | 33 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 34 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
  Spain | 7 | 8 | 15
  Taiwan | 10 | 9 | 19
  Lithuania | 2 | 2 | 4
  Israel | 3 | 4 | 7
  India | 2 | 1 | 3
  Canada | 3 | 1 | 4
  Denmark | 1 | 1 | 2
  Australia | 1 | 0 | 1
  Latvia | 2 | 3 | 5
  Japan | 14 | 15 | 29
  New Zealand | 5 | 6 | 11
  Korea, Republic of | 9 | 9 | 18
  Sweden | 0 | 1 | 1
Surgical screw type [Number; unit: participants] — Surgical screws used in initial surgery to repair femur neck hip fracture.
  participants
    Cancellous Screws | 54 | 53 | 107
    Sliding Hip Screws | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Revision Surgery at 12 Months After Internal Fixation of a Low-Trauma Femoral Neck Fracture
Description: Revision surgery (re-operation) was defined as any additional surgical intervention performed or recommended at the site of the index procedure, except those that were planned at the time of the index procedure.
Time Frame: 12 months
Population: Participants who were randomized and received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 60 | 61
percentage of participants | 87 [77 to 93] | 86 [76 to 92]

2. Secondary Outcome: Percentage of Participants With Radiographic Evidence of Healing
Description: The signs of femoral neck fracture healing included disappearance of the fracture line on radiographs. If a participant had radiographic evidence of healing at the 12-month visit, that participant was considered to have radiographic evidence of healing.
  Percentage was calculated as: (number of participants with radiographic evidence of healing / total number of participants analyzed) * 100.
Time Frame: Randomization up to 12 months
Population: Participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 60 | 61
percentage of participants | 78.3 | 78.7

3. Secondary Outcome: Percentage of Participants With Pain Control During Ambulation
Description: The worst pain numeric rating scale (NRS) was used to assess the impact of pain on a participant's life. NRS Item 3 assessed the worst musculoskeletal pain severity during the walking test. Pain was measured by an 11-point Likert scale. The following cut-points were used to categorize the NRS responses: 0 = no pain, 1 to 4 = mild pain, 5 to 6 = moderate pain, and 7 to 10 = severe pain. Participants with an NRS score of <7 were categorized as having no severe fracture-site pain with ambulation and no worsening of NRS scores >2 from baseline. Percentage was calculated as: (Number of participants with pain control during ambulation / total number of participants) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received treatment, and had baseline and at least one nonmissing post-baseline measurement. Last observation carried forward (LOCF) values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 47 | 49
percentage of participants | 91.5 | 89.8

4. Secondary Outcome: Percentage of Participants Without Severe Fracture-Site Pain During 24 Hours Prior to Visit
Description: The worst pain NRS was used to assess the impact of pain on a participant's life. Fracture-site pain severity was assessed for pain in the 24 hours preceding a visit. Pain was measured by an 11-point Likert scale. Participants with an NRS score of <7 in the 24 hours preceding a visit and no worsening of NRS >2 from baseline were categorized as having no severe fracture-site pain. Percentage was calculated as: (number of participants with pain control during 24 hours preceding a visit / total number of participants) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug and had baseline and at least one nonmissing post-baseline measurement for severe fracture-site pain in the last 24 hours. LOCF values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 50 | 51
percentage of participants | 88.0 | 82.4

5. Secondary Outcome: Percentage of Participants Without Severe Fracture-Site Pain During Weight Bearing
Description: The worst pain NRS was used to assess the impact of pain on a participant's life. Fracture-site pain severity was assessed for pain on weight bearing. Pain was measured by an 11-point Likert scale. Participants with an NRS score of <7 during weight bearing and no worsening of NRS >2 from baseline were categorized as having no severe fracture-site pain. Percentage was calculated as: (number of participants with pain control during weight bearing / total number of participants) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug and had baseline and at least 1 nonmissing post-baseline measurement. LOCF values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 47 | 50
percentage of participants | 89.4 | 88.0

6. Secondary Outcome: Percentage of Participants With Functional Evidence of Healing
Description: Functional healing was defined as ability to walk with a gait speed ≥ 0.05 meters/second (m/s) with a change from baseline ≥ -0.1 m/s. The walking test involved having the participant walk a distance of 7 meters (m) at a self-selected, comfortable pace. A 4-m portion of the test was timed to determine the participant's gait speed in m/s.
  Percentage was calculated as: (number of participants with functional evidence of healing / total number of participants analyzed) * 100.
Time Frame: 12 Months
Population: Participants who were randomized, received at least 1 dose of study drug, and had either at least one nonmissing gait speed or non-ambulatory status. LOCF values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 48 | 50
percentage of participants | 85.4 | 74.0

7. Secondary Outcome: Percentage of Participants Able to Ambulate
Description: Ability to ambulate was defined as ambulatory with convalescent aid or without convalescent aid. Percentage was calculated as: (number of participants able to ambulate / number of total participants analyzed) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized and received at least 1 dose of study drug and had at least 1 nonmissing post-baseline measurement. LOCF values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 48 | 50
percentage of participants | 97.9 | 98

8. Secondary Outcome: Percentage of Participants Who Regain Their Prefracture Ambulatory Status
Description: Prefracture ambulatory status was defined as either ambulatory with or without a walking aid. A participant was considered to have regained their prefracture ambulatory status if the participant's postsurgery ambulatory status was returned to or was improved from their pre-surgery ambulatory status. Percentage was calculated as = (number of participants who regained their ambulatory status / total number analyzed) * 100.
Time Frame: Up to 12 months
Population: Participants who were randomized, received at least 1 dose of study drug, and had baseline and at least one nonmissing post-baseline measurement. LOCF values used.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 56 | 58
percentage of participants | 73.2 | 56.9

9. Secondary Outcome: Mean Change From Baseline to 6 Months in Worst Fracture-Site Pain
Description: The worst pain NRS was used to assess the impact of pain on a participant's life. Participants with an NRS score of <7 were categorized as having no severe fracture-site pain. Least Squares (LS) means was calculated using analysis of covariance (ANCOVA) and adjusted for baseline, treatment group, region, fracture type, and fixation type.
Time Frame: Baseline, 6 Months
Population: Participants who were randomized and received at least 1 dose of study drug and had baseline and at least 1 nonmissing post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 47 | 50
units on a scale
  During ambulation (n = 45, 46) | 0.2 (0.37) | 0.2 (0.36)
  During 24 hours preceding visit (n = 47, 50) | -0.3 (0.45) | -0.8 (0.42)
  On weight bearing (n = 46, 49) | 0.7 (0.39) | 0.8 (0.36)

10. Secondary Outcome: Mean Change From Baseline to 6 Months in Gait Speed
Description: The walking test involved having the participant walk a distance of 7 m at a self-selected, comfortable pace. A 4-m portion of the test was timed to determine the participant's gait speed in m/s. LS means was calculated using ANCOVA and adjusted for baseline, treatment group, region, fracture type, and fixation type.
Time Frame: Baseline, up to 6 Months
Population: Participants who were randomized, received at least 1 dose of study drug and had baseline and at least one nonmissing post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 45 | 47
m/s | -0.672 (2.128) | 1.524 (2.018)

11. Secondary Outcome: Time to Revision Surgery
Description: Time to revision surgery was defined as the time from initial hip fracture surgery to revision surgery, or recommendation for revision surgery if recommended but not performed. Time to revision surgery was censored at the date of the last contact.
Time Frame: Baseline to revision surgery (up to 14.14 Months)
Population: Participants who were randomized, received at least 1 dose of study drug, and who did not have revision surgery or if they had revision surgery, it was adjudicated as not being related to the initial hip fracture surgery. Participants censored: Teriparatide = 51; placebo = 51.
Measure: Median (Full Range); unit: days
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 60 | 59
days | 358.5 [15 to 430] | 350 [12 to 412]

12. Secondary Outcome: Mean Change From Baseline to 6 Months on Short Form-12 (SF-12) Physical (PCS) and Mental Component Summary (MCS) Scores
Description: SF-12 is a self-reported questionnaire covering a mental component score (MCS) and a physical component score (PCS), each scoring from a 0 to 100 (worst to best) scale. LS mean was calculated using ANCOVA and adjusted for baseline, treatment group, region, fracture type, fixation type, visit, and visit-by-treatment interaction.
Time Frame: Baseline, up to 6 Months
Population: Participants who were randomized, received at least 1 dose of study drug, were adjudicated as having the hip fracture in the neck of the femur and had baseline and at least 1 nonmissing post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale
  PCS Month 6 (n = 49, 49) | -3.73 (1.2) | -4.75 (1.2)
  MCS Month 6 (n = 49, 49) | -0.58 (2.1) | -0.49 (2.1)

13. Secondary Outcome: Mean Change From Baseline to 6 Months on Western Ontario McMaster Osteoarthritis Index (WOMAC)
Description: WOMAC is: a self-reported questionnaire that consisted of 24 questions covering 3 health domains: Pain (5 items: during walking, using stairs, in bed, sitting or lying, and standing), Stiffness (2 items: after first waking and later in the day), and Physical Function. Each domain was scored by summing the individual items and transforming the scores into a 0 to 100 (best to worst) scale. LS mean was calculated using ANCOVA and adjusted for baseline, treatment group, region, fracture type, fixation type, visit, and visit-by-treatment interaction.
Time Frame: Baseline, up to 6 Months
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 58 | 59
units on a scale
  Physical Function Score - Month 6 (n=48, 51) | 12.9 (4.36) | 12.8 (4.25)
  Pain Score - Month 6 ( n = 51, 51) | 8.2 (3.76) | 10.3 (3.68)
  Stiffness Score - Month 6 (n = 51, 51) | 13.1 (3.78) | 11.8 (3.75)

14. Secondary Outcome: Mean Change From Baseline to 6 Months on European Quality of Life Questionnaire (EQ-5D) Health State Score
Description: The EQ-5D is a 5-item, self-reported, generic, multidimensional, health-related, quality-of-life instrument with 5 items. Overall health state score was also self-reported using a visual analogue scale (VAS) marked on a scale scored from 0 (worse imaginable health state) to 100 (best imaginable health state). LS mean was calculated using ANCOVA and adjusted for baseline, treatment group, and region.
Time Frame: Baseline, up to 6 Months
Population: All randomized participants who were randomized, received at least 1 dose of study drug, were adjudicated as having the hip fracture in the neck of the femur, and had baseline and at least 1 nonmissing post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Placebo
Number analyzed (Participants) | 51 | 51
units on a scale | 7.4 (4.02) | 7.6 (3.87)

ADVERSE EVENTS:
Time Frame: Randomization to Study Completion
Groups:
- Placebo Follow-up: Follow-up after placebo once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
- Teriparatide Follow-up: Follow-up after teriparatide 20 µg once-daily by SC injection for 6 months. Participants received calcium and vitamin D supplements.
Arm/Group | Placebo | Teriparatide | Placebo Follow-up | Teriparatide Follow-up
Serious Adverse Events (participants affected / at risk) | 6/61 | 2/60 | 6/53 | 2/49
Other Adverse Events (participants affected / at risk) | 34/61 | 31/60 | 18/53 | 16/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=61) | Teriparatide (N=60) | Placebo Follow-up (N=53) | Teriparatide Follow-up (N=49)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=61) | Teriparatide (N=60) | Placebo Follow-up (N=53) | Teriparatide Follow-up (N=49)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Periodontal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sense of oppression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0/44 (0) | 0/43 (0) | 1/39 (1) | 0/39 (0)
Prostatitis (Reproductive system and breast disorders) | 0/17 (0) | 1/17 (1) | 0/14 (0) | 0/10 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/44 (1) | 0/43 (0) | 0/39 (0) | 0/39 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sebaceous cyst excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days